CLINICAL TRIAL: NCT06116149
Title: Strategies for Implementing a Postpartum Lifestyle Intervention in WIC Clinics: A Cluster Randomized Trial
Brief Title: Strategies for Implementing a Postpartum Lifestyle Intervention in WIC Clinics
Acronym: STRIVE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Tulane University (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH); Pennington Biomedical Research Center (Other); University of Pennsylvania (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2022-1294; OT2HL158287 (NIH)
Record Dates: First submitted 2023-09-29; First posted 2023-11-03 (Actual); Last update posted 2025-07-25 (Actual); Status verified 2025-07

CONDITIONS: Obesity; Gestational Diabetes; Lifestyle, Healthy; Glucose Intolerance During Pregnancy; PreDiabetes; Hyperglycemia
Keywords: Diabetes Prevention Program
MeSH Terms: conditions — Obesity; Diabetes, Gestational; Prediabetic State; Hyperglycemia

STUDY DESIGN:
Intervention Model Description: Cluster-randomization of 38 Women, Infants, and Children (WIC) clinics
Masking Description: Due to the nature of the cluster design and intervention program, the study participants, health coaches, DPP Coordinators, WIC clinic staff, and research staff who collect clinical outcome data will not be blinded.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- In-person health coach strategy (Active Comparator): Delivery of 24 health coaching sessions in-person by health coaches over 1 year.
  Standard delivery of 24-sessions of the Group Lifestyle Balance (GLB) behavioral intervention in WIC clinics. The GLB was adapted from the original Lifestyle Balance behavioral intervention used in the original Diabetes Prevention Program trial for use in community translation and group settings. It focuses on improving diet and physical activity and promoting moderate weight loss through health coaching on behavioral change, including self-monitoring of food intake, physical activity, and weight.
  Interventions: Behavioral: In-person health coach delivery of the GLB
- Multifaceted technology-assisted health coach implementation strategy (Active Comparator): Delivery of 12 health coaching GLB sessions in-person by health coaches over one year; supplemental technology support, including tools for self-monitoring, health coach monitoring, asynchronous delivery of intervention materials, and asynchronous coach and group connection.
  The GLB was adapted from the original Lifestyle Balance behavioral intervention used in the original Diabetes Prevention Program trial for use in community translation and group settings. It focuses on improving diet and physical activity and promoting moderate weight loss through health coaching on behavioral change, including self-monitoring of food intake, physical activity, and weight.
  Interventions: Behavioral: Technology-assisted health coach delivery of the GLB

INTERVENTIONS:
Behavioral: In-person health coach delivery of the GLB — Delivery of 24 health coaching sessions in-person by health coaches over 1 year.
  Standard delivery of 24-sessions of the Group Lifestyle Balance (GLB) behavioral intervention in WIC clinics. The GLB was adapted from the original Lifestyle Balance behavioral intervention used in the original Diabetes Prevention Program trial for use in community translation and group settings. It focuses on improving diet and physical activity and promoting moderate weight loss through health coaching on behavioral change, including self-monitoring of food intake, physical activity, and weight.
  Arms: In-person health coach strategy
Behavioral: Technology-assisted health coach delivery of the GLB — Delivery of 12 health coaching GLB sessions in-person by health coaches over one year; supplemental technology support, including tools for self-monitoring, health coach monitoring, asynchronous delivery of intervention materials, and asynchronous coach and group connection.
  The GLB was adapted from the original Lifestyle Balance behavioral intervention used in the original Diabetes Prevention Program trial for use in community translation and group settings. It focuses on improving diet and physical activity and promoting moderate weight loss through health coaching on behavioral change, including self-monitoring of food intake, physical activity, and weight.
  Arms: Multifaceted technology-assisted health coach implementation strategy

SUMMARY:
The primary objective of the STRIVE study is to compare two implementation strategies for Diabetes Prevention Program delivery: an in-person health coach strategy (standard 24 in-person sessions at WIC clinics) vs. a multifaceted technology-assisted health coach implementation strategy (12 in-person sessions at WIC clinics supplemented by technology support) on implementation and health-related outcomes in postpartum women.

DETAILED DESCRIPTION:
The overall objective of this project is to study the implementation, effectiveness, and sustainability of implementing the Diabetes Prevention Program (DPP) in postpartum women who receive services from WIC. In this effectiveness-implementation type III cluster-randomized trial, we will compare two implementation strategies for DPP delivery: an in-person health coach-led implementation strategy (standard 24 in-person sessions) vs. a multifaceted technology-assisted health coach implementation strategy (12 in-person sessions supplemented by technology tools).

Nineteen clinics will be randomized to the multifaceted technology-assisted health coach strategy and 19 to the in-person health coach-led strategy. A total of 722 postpartum participants (19 per clinic) will be recruited into the study and followed for 12 months for implementation and effectiveness outcomes. A post-intervention study visit will take place 6 months after the end of the 12-month intervention to evaluate the sustainability of the implementation strategies.

ELIGIBILITY:
Inclusion Criteria for Clinics:

* Serve a large number of WIC postpartum participants
* Willing and able to provide space for the study

Inclusion Criteria for Participants:

* Age 18 or older
* Gave birth in the past 6 weeks to 12 months
* Obesity or history of gestational diabetes mellitus (Current BMI ≥30 kg/m², OR Medical-record documented history of gestational diabetes mellitus and BMI ≥25 kg/m²)
* No self-reported diabetes (other than gestational diabetes)
* Hemoglobin A1c <6.5%
* Not currently pregnant or planning to become pregnant in the next 6 months
* No plans to move outside of the study region in the next 12 months
* Access to a smartphone
* Willing and able to participate in the intervention and provide consent
* Not an immediate family member of the staff at the WIC clinic
* Other concerns regarding ability to meet trial requirements, at the discretion of the principal investigator or study coordinator

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 722 (Estimated)
Dates: Start 2023-12-12 (Actual); Primary Completion 2026-10 (Estimated); Study Completion 2027-04 (Estimated)

PRIMARY OUTCOMES:
Difference in uptake (primary implementation outcome) | Measured from baseline to 12 months
  The primary implementation outcome will be the difference between study arms in a composite uptake score, as defined by a composite score consisting of the percent of sessions attended and the percentage of times in which participants record weight, activity, and diet compared to what is recommended by the intervention.
Difference in mean 12-month weight reduction (primary health-related outcome) | Measured at 3, 6, 9 and 12 months
  The primary health-related outcome will be difference in mean weight reduction from baseline to 12 months between study arms

SECONDARY OUTCOMES:
Fidelity | 12 months
  Percentage of sessions held
Acceptability | Measured at baseline, 6, and 12 months
  Acceptability scores for participants, DPP coordinators, DPP coaches, WIC clinic management. Measured by survey; higher score means better outcome.
Appropriateness | baseline
  Appropriateness scores for participants, DPP coordinators, DPP coaches, WIC clinic management. Measured by survey; higher score means better outcome.
Feasibility (suitability) | Baseline
  Feasibility scores for participants, DPP coordinators, DPP coaches, and WIC clinic management. Measured by survey; higher score means better outcome.
Adoption (WIC clinics) | Baseline
  Percentage of invited WIC clinics adopting the DPP program. Measured by study administrative data.
Adoption (WIC nutritionists) | Baseline
  Percentage of invited WIC nutritionists being trained. Measured by study administrative data.
Adoption (WIC health educators) | Baseline
  Percentage of invited WIC health educators being trained. Measured by study administrative data.
Penetrance (participants) | 12 months
  Percentage of enrolled participants receiving assigned intervention. Measured by study administrative data.
Penetrance (WIC DPP coordinators) | 12 months
  Percentage of percentage of trained WIC DPP coordinators supporting health coaches. Measured by study administrative data.
Penetrance (WIC health coaches) | 12 months
  Percentage of percentage of trained WIC DPP health coaches delivering the intervention. Measured by study administrative data.
Percentage of participants who were either eligible, screened, or contacted who were enrolled. | Baseline
  Reach
Cost-effectiveness | 12 months
  Incremental direct costs (intervention) per additional percentage of individuals reaching weight loss goal at 12 months
Difference in mean 12-month change in percent weight reduction | Measured from baseline to 12 months
  Difference in mean percent weight reduction from baseline to 12 months between study arms
Difference in mean 12-month change in physical activity | Measured from baseline to 12 months
  Difference in mean change in physical activity from baseline to 12 months between study arms, as assessed by metabolic equivalent (MET)-h/week (measured by validated questionnaire)
Difference in mean 12-month change in healthy eating index | Measured from baseline to 12 months
  Difference in mean change in healthy eating index from baseline to 12 months between study arms, as assessed by 24-hour dietary recalls (range 0 to 100; higher scores mean healthier eating pattern)
Difference in mean 12-month change in waist circumference | Measured from baseline to 12 months
  Difference in mean change in waist circumference from baseline to 12 months between study arms
Difference in mean 12-month change in hemoglobin A1c | Measured from baseline to 12 months
  Difference in mean change in hemoglobin A1c from baseline to 12 months between study arms
Difference in mean 12-month change in systolic blood pressure | Measured from baseline to 12 months
  Difference in mean change in systolic blood pressure from baseline to 12 months between study arms
Difference in mean 12-month change in diastolic blood pressure | Measured from baseline to 12 months
  Difference in mean change in diastolic blood pressure from baseline to 12 months between study arms
Difference in mean 12-month change in health-related quality of life (HRQoL) | Measured from baseline to 12 months
  Difference in mean change in health-related quality of life (HRQoL) from baseline to 12 months between study arms (assessed by short form (SF)-12, validated survey)
Difference in proportion of participants meeting intervention goals at 12 months | Measured from baseline to 12 months
  Assessed by validated questionnaires, 24-hour dietary recalls, and weight measurements

OTHER OUTCOMES:
Sustainability (DPP coordinators): comparison of perceived sustainability of the two implementation strategies among WIC staff | 18 months
  Assessed by surveys and interviews
Sustainability (Participants): comparison of the proportion of participants maintaining DPP goals at six months after their participation in the DPP has ended | 18 months
  Assessed by validated questionnaires, 24-hour dietary recalls, and weight measurements

CONTACTS AND LOCATIONS:
Locations (1):
- Tulane University School of Public Health and Tropical Medicine, New Orleans, Louisiana, United States

IPD SHARING:
Plan to Share IPD: Yes
Our study data sharing plan will comply with all NIH policies for data sharing. Data sharing will be implemented in a timely manner. Study data, including data from baseline and follow-up visits, will be prepared sharing. Data will be prepared by the study data manager/biostatistician. These data will be free of identifiers that allow identification of individual research participants either directly or through "deductive disclosure." We are very open to sharing data enthusiastically with the general scientific community, since we also believe in the added value of other investigators working on these data.
Supporting Information: Study Protocol, SAP
Time Frame: Data sets will be prepared for sharing no later than 3 years after the end of the final patient follow-up visit or 2 years after the main paper of the trial has been published, whichever comes first.
Access Criteria: We will offer opportunities for outside investigators to collaborate with us using complete study data.